CLINICAL TRIAL: NCT05387031
Title: Efficacy of Ustekinumab-based Integrated Medicine Therapy in Patients With Symptomatic Stricturing Crohn's Disease: a Multicenter, Prospective, Observational Cohort Study
Brief Title: Efficacy of Ustekinumab Therapy in Patients With Symptomatic Stricturing Crohn's Disease
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Second Affiliated Hospital of Soochow University (Other); Chongqing Renji Hospital, University of Chinese Academy of Sciences (Other Government); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Seventh Medical Center of PLA Army General Hospital (Other); First People's Hospital of Hangzhou (Other); Yangzhou University (Other); Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-0276
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease; Stricture; Bowel; Intestinal Stricture
Keywords: Crohn Disease; intestinal stricture; Ustekinumab; integrated medicine therapy; cohort study
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed tissue，blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with symptomatic stricturing Crohn's disease: The decision to start ustekinumab was at the discretion of the treating physician. The initial intravenous (IV) infusion with ustekinumab at baseline was weight-adjusted (260 mg ≤55 kg, 390 mg between 55 and 85 kg, 520 mg ≥85 kg). According to the label, the first subcutaneous (SC) 90 mg induction dose was administered at week 8 followed by a maintenance dose of 90 mg SC every 8 or 12 weeks, at the discretion of the physician.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — The initial intravenous (IV) infusion with ustekinumab at baseline was weight-adjusted (260 mg ≤55 kg, 390 mg between 55 and 85 kg, 520 mg ≥85 kg). According to the label, the first subcutaneous (SC) 90 mg induction dose was administered at week 8 followed by a maintenance dose of 90 mg SC every 8 or 12 weeks, at the discretion of the physician. This study evaluated the CD disease activity, obstructive symptoms, and radiographic or endoscopic remission in patients at different follow-up time points, and comprehensively evaluated the efficacy of ustekinumab in relieving stenotic CD and its related factors.
  Other Names: Stelara

SUMMARY:
This study intends to select patients with confirmed moderate-to-severe Crohn's disease (CD) and obstructive symptoms of intestinal stenosis, who have clear evidence of lumen stenosis caused by the disease itself through radiography or endoscopy. After the informed consent of the patients, comprehensive drug therapy with ustekinumab as the mainstay was performed. The basic information and medical history of the patients were collected, and the treatment process of the patients was followed up and recorded, and the drug regimen was adjusted according to the physician's experience and judgment. At different follow-up time points, blood, feces, tissue and other specimens of patients were collected according to the situation, and gastrointestinal endoscopy, imaging examination, laboratory index examination, self-assessment of subjects' symptoms, and nutritional risk screening were performed on the patients. This study evaluated the CD disease activity, obstructive symptoms, and radiographic or endoscopic remission in patients at different follow-up time points, and comprehensively evaluated the efficacy of ustekinumab in relieving stenotic CD and its related factors.

DETAILED DESCRIPTION:
This study intends to select patients with confirmed moderate-to-severe CD and obstructive symptoms of intestinal stenosis, who have clear evidence of lumen stenosis caused by the disease itself through radiography or endoscopy. After the informed consent of the patients, comprehensive drug therapy with ustekinumab as the mainstay was performed. The basic information and medical history of the patients were collected, and the treatment process of the patients was followed up and recorded, and the drug regimen was adjusted according to the physician's experience and judgment. At different follow-up time points, blood, feces, tissue and other specimens of patients were collected according to the situation, and gastrointestinal endoscopy, imaging examination, laboratory index examination, self-assessment of subjects' symptoms, and nutritional risk screening were performed on the patients. This study evaluated the CD disease activity, obstructive symptoms, and radiographic or endoscopic remission in patients at different follow-up time points, and comprehensively evaluated the efficacy of ustekinumab in relieving stenotic CD and its related factors.

The investigators conduct follow-up and disease assessment at weeks 0, 12, 24, 52, and 104, respectively. The investigators define the primary endpoint of the study as the treatment success of ustekinumab at week 52, and investigate the efficacy of ustekinumab by site of stricture and assessed possible clinical, biochemical, and radiological predictors of treatment response at weeks 12, 24, 52, and 104. This clinical study provides evidence for the efficacy of ustekinumab-based comprehensive drugs in the treatment of stenotic Crohn's disease, provides biological information resources for future treatment options for patients with stenotic CD, and can also be used for disease diagnosis and treatment. In this group of people, the investigators tend to further analyze and find the influencing factors related to the development of stenotic CD disease and drug response, in order to provide corresponding support for clinical activities in the early stage of the disease or during the treatment process, and to improve the effectiveness and accuracy of individualized treatment for patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe Crohn's disease
* Obstructive symptoms within the last eight weeks
* A single or several lumen stricture(s) identified by radiological imaging or endoscopy
* For strictures identified by CT enterograph defined as a lesion with combination of a reduction of luminal narrowing >50%, an increase in bowel wall thickness >25% relative to non-affected bowel and pre-stricture dilation >3.0 cm
* For strictures identified during endoscopic procedure defined by intestinal strictures with a lumen diameter ≤12 mm or even inability to pass the endoscope across the narrowing

Exclusion Criteria:

* Requirement of urgent surgery or endoscopic intervention within 2 months as judged by the clinician
* Symptoms or signs of perforation such as active perianal sepsis, abdominal abscess, intestinal fistula, and abdominal adhesions
* Intestinal obstruction caused by surgery, intra-abdominal abscess, isolated intestinal stricture
* Effective treatments for stricture in the past half a year, such as endoscopic balloon dilatation, intestinal stricture plasty, surgery/manual anal dilatation, etc.
* Unable to eat after using enteral nutrition for more than 2 months
* History of ustekinumab (UST) or other IL-23 antagonists use in the past 12 months
* CT enterograph contraindications, such as allergy to contrast media
* Relative contraindications of biological agents, such as pulmonary tuberculosis-positive chest X-ray or active tuberculosis with strong positive tuberculin skin test, myocardial infarction, heart failure, or demyelinating neurological disease
* Currently suffering from a solid tumor, lymphoma, or melanoma and undergoing chemotherapy or radiation therapy
* Combination of intestinal dysplasia (eg, diagnosed with short bowel syndrome), colostomy, or colorectal tumors
* Combination of active gastrointestinal bleeding, shock, severe diarrhea, refractory vomiting and severe malabsorption syndrome
* Combination of severe liver and kidney dysfunction
* Coexistence of bacterial or viral active infection
* Pregnant or breastfeeding
* Severe hemodynamics, unstable vital signs or presence of rapidly progressive or end-stage disease, expected to be fatal during the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were adult CD patients treated with their first UST therapy for symptomatic strictures (confirmed on endoscopy or imaging) from centers of IBD at 8 hospitals all over China. This study does not involve the use of vulnerable groups.
Sampling Method: Probability Sample
Enrollment: 239 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment success at week 52 | up to 52 weeks
  The primary endpoint was the success at week 52, defined as ustekinumab continuation with all the following criteria: (1) no use of a prohibited treatment (corticosteroids after the eight week following inclusion, parenteral nutrition, other biological agents); (2) no endoscopic dilation; (3) no bowel surgery for resection of small bowel stricture; (4) no severe adverse events leading to ustekinumab withdrawal and (5) no study withdrawal whatever the reason.
  Clinical improvement was measured by symptoms and clinical remission (Crohn's Disease Activity Index <150), steroid-free symptom improvement (obstructive symptom score) following initial steroid tapering, Crohn's Disease Obstructive Score (improvement of ≥1 point), treatment failure (defined as bowel obstruction requiring surgery, endoscopic balloon dilation, or persisting symptoms necessitating change in treatment), the need for surgery.

SECONDARY OUTCOMES:
Number of participants with improvement in stricture inflammation and morphology on imaging | at week 8, 24, 52 and 104
  CT and MRI stricture improvement was defined as resolution of prestenotic dilatation (small bowel diameter <3.0 cm); stricture resolution (normal bowel wall thickness and luminal diameter with absence of prestenotic dilation; and reduced stricture length by ≥1 mm). Intestinal ultrasound stricture improvement included normalisation of prestenotic dilation (<3.0 cm) or reduction in prestenotic dilation (≥50%). Endoscopic stricture improvement included increased luminal diameter; the ability to pass a standard paediatric colonoscope (11.5 mm diameter); and improved stricture ulceration score using SES-CD or DBE-CD.
Number of participants with improvement in general health | at week 8, 24, 52 and 104
  General health improvement was measured by patient reported outcomes of Inflammatory Bowel Disease (IBD) Quality of Life Questionnaire. The minimum and maximum values are 32 and 224 points respectively, and higher scores mean a better outcome.
Number of Participants with surgery | at week 8, 24, 52 and 104
  Number of Participants with surgery during follow-up included patients undergoing any surgery for endoscopic dilatation and stricture resection.
Number of participants with treatment success at week 104 | at week 104
  Success at week 104 was defined in the same way as in week 52.

OTHER OUTCOMES:
Clinical response and clinical alleviate | at week 8, 24, 52 and 104
  Clinical response was defined as HBI reduce at least three points, alleviate clinical alleviate defined as HBI ≤ 4 points, CDAI < 150 points.
Biochemical ease | at week 8, 24, 52 and 104
  Fecal calprotectin (FC) level ≤ 200 μg/g and/or CRP≤5 mg/L, or decrease ≥ 50%, compared to the baseline significant.
UST drug concentration and antibody concentration | at week 8, 24, 52 and 104
  Measurements of UST drug concentration and antibody concentration, and their relationship with improvement of inflammation or imaging (CT enterography, bowel ultrasound, and endoscopy).
Safety outcomes | at week 8, 24, 52 and 104
  Safety outcomes included the number of drug-related adverse events, infections, and disease-related hospitalizations per 100 patients per year. Adverse events were categorized as: possibly related, probably related, and not related to UST. Infections were classified as: 1) mild: infections that did not require medication; 2) moderate: infection treated with oral antibiotics or antiviral drugs; (3) Severe: infection requiring hospitalization or treatment with intravenous antibiotics or antiviral drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, MD., Study Chair — Center of IBD, the Second Affiliated Hospital, Zhejiang University School of Medicine; Jingwen Liu, MD., Principal Investigator — Center of IBD, the Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (8):
- China (8):
  - Department of Gastroenterology, Seventh Medical Center of PLA Army General Hospital, Beijing, Beijing Municipality
  - Department of Gastroenterology, Chongqing Renji Hospital, University of Chinese Academy of Sciences, Chongqing, Chongqing Municipality
  - Department of Gastroenterology, Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Gastroenterology, Huai'an First People's Hospital, Huai'an, Jiangsu
  - Department of Gastroenterology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Department of Gastroenterology, Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Center of Inflammatory Bowel Disease, Department of Gastroenterology, the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Department of Gastroenterology, The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang